CLINICAL TRIAL: NCT04473755
Title: A Naturalistic Study of Functional Impairment for Individuals With ADHD in the Early Morning and Late Afternoon/Evening Hours
Status: Completed | Type: Observational
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Other Study IDs: 800012103
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; impairment; symptoms
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD: This group will include participants who meet DSM-5 diagnostic criteria for ADHD and meet all other study inclusion criteria.
- Non-ADHD: This group will include participants who do not meet DSM-5 diagnostic criteria for ADHD and meet all other study inclusion criteria.

SUMMARY:
The objective of this study is to assess the burden and impact of ADHD impairment in the early morning and late afternoon/evening hours for adolescents and young adults. Functional impairments will focus on the currently identified areas of functional impairment in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5, American Psychiatric Association, 2013) - namely, social, academic, and occupational functioning. This is necessary for two reasons: (1) the current literature on ADHD impairment and functioning is concentrated within elementary school children; and (2) studies of intervention effectiveness are typically concentrated during the school day. This current state of the literature ignores the obvious - as ADHD is a chronic disorder, it needs to be addressed as children grow into adolescence and young adulthood, and it needs to be remediated at times outside of the school day such as in the morning and late afternoon/evening.

Therefore, the specific areas assessed in the present study will relate to driving, school, work, and family functioning. These are important areas to study, as the research literature has typically focused on elementary school and school-day behavior in assessments of symptom presentation, impairment, and treatment outcome. As individuals with ADHD grow older, the entire day becomes relevant in determinations of functioning (e.g., workdays may begin in the very early morning or last into the evening/night), and productivity can be assessed across waking hours rather than just across the elementary school day. Once areas of functional impairment in these times of day are determined, for this age group, treatment candidates can aim to address these treatment targets.

DETAILED DESCRIPTION:
Study aims are as follows:

1. To investigate the impairment present in the morning and late afternoon/evening for individuals with ADHD, relative to a non-ADHD group.

   a. Hypothesis: Individuals with ADHD will illustrate more impaired functioning in the morning and late afternoon/evening, relative to a non-ADHD group in the following domains: i. Risky Driving ii. School/Workplace related behavior (e.g., time on-task in the evening, management of weekly schedule) iii. Family and social functioning
2. Develop a set of recommendations for the evidence-based assessment of morning and late afternoon/evening behavior of individuals with ADHD.

   1. Hypothesis: It is hypothesized that a multi-method, multi-domain assessment of impaired functioning will yield the most clinically defensible assessment approach.

Rolling enrollment will be used in this study. Participants will attend an intake visit to provide informed consent for participation in the study, and collect baseline and diagnostic information. The targeted population will be youth and young adults between the ages of 16-30 with a valid driver permit or license. To determine eligibility for the study, participants will complete (1) a self-report of ADHD symptoms (Molina, Smith, & Pelham, 2001; Pelham, Gnagy, Greenslade, & Milich, 1992), (2) the Impairment Rating Scale (Fabiano et al., 2006; Sibley et al., 2012a); and (3) a semi-structured Disruptive Behavior Disorders interview with a clinician to obtain contextual information on symptoms and impairment over the last six months (Hartung et al, 2005). Participants will also complete the WASI-2 to ascertain an estimate of IQ. Additionally, a collateral rater (i.e., parent or significant other; Sibley et al., 2012a, 2012b) will report on the participant's ADHD symptom ratings for the past six months and retrospectively provide a report on childhood symptoms. The collateral rater will also complete an Impairment Rating Scale based on the last six months. Participants will be classified as ADHD if there are at least 4 symptoms of inattentive and/or hyperactive-impulsive behaviors endorsed at clinically significant levels, evidence of onset of ADHD prior to age 12, and current psychosocial impairment (Sibley et al., 2012a, 2012b).

To reduce variability between the ADHD and non-ADHD groups, we will match participants on age (+/- 2 years), sex, and whether they are employed or unemployed.

Eligible participants in either the ADHD or non-ADHD group will then have a meeting with the research team to initiate data collection methods over a two-week time period (i.e., 14 early morning and 14 late afternoon/evening assessments; N=28 assessments/participant total). This amount of repeated measurement should be adequate for detecting differences in participants (e.g., Ferguson et al., 2012). To accurately capture the diverse array of potential functional impairments in the early morning and late afternoon/evening hours, a multi-method approach to data collection will be utilized. The keystone of the data collection process will be via the adolescent/young adult's smart phone. In our data collection approach we will use commercially available and commonly employed (e.g., smartphones) measurement tools to develop a method of data collection that may be eventually appropriate for scale in the adolescent/young adult population. Using an application that permits geo-location, information on driving, and timestamps for location (e.g., Life360.com), the participants' self-management within key functional domains will be assessed. The following data will be collected:

Morning and Evening Routine. Participants will provide a weekly schedule for the upcoming week. Using this information, mobile technology will be used to determine success with meeting expectations for morning routine (e.g., waking up; leaving for school/work; falling asleep). Mobile technology will track sleeping habit and time of wakening, and geo-fencing will set an alert when the participant leaves the home. Using an idiographic list of responsibilities for work/school/home, we will monitor performance toward goal attainment as we have done in related studies in the natural and laboratory setting (Fabiano et al., 2010; Fabiano et al., 2018).

Driving. Early morning and late afternoon/evening driving will be monitored using the participants' smartphone application, which includes the Driver Protect feature. Driver Protect includes driving reports that include potentially unsafe behaviors (phone use to text while driving, speeding, hard braking, collisions) as well as 30 days of location history. We will collect companion driving performance information using the Life360 app which will log all trips conducted by the driver, total miles traveled, record top speed for each trip, and record frequency counts of hard/extreme braking and acceleration. Similar tools have been successfully used in prior studies (Fabiano et al., 2011; Fabiano et al., 2016) and they are well-tolerated by participants.

Family and Social Functioning. Ecological, momentary assessment will be used to assess family and social functioning based on report from both the participant and identified collateral(s). Ecological, momentary assessment is an approach that uses a smartphone based prompt (i.e., in a text message) to ask the participant about behavior/functioning/mood at that moment (e.g., Miguelez-Fernandez, et al., 2018). Participants and collaterals will be contacted in the early morning and late afternoon/evening hours to obtain information on typical activities, individuals they are interacting with, and to obtain a brief rating of functional impairment using the Impairment Rating Scale (Fabiano et al., 2006). Participants and collaterals will be contacted at least once each morning and once each afternoon/evening daily, for two weeks.

ADHD Symptoms and Impairment. As part of the assessment of family and social functioning probes, we will also administer a brief probe of ADHD symptoms and impairment. We will include the six symptoms from the Adult ADHD Self-Report Scale (Kessler, et al., 2007) and the overall impairment item on the Impairment Rating Scale (Fabiano et al., 2006). Data for this measure will be collected during both the early morning and late afternoon/evening assessment periods.

Our prior work illustrated little reactivity with observations of behavior, even in high-profile situations such as driving. Indeed, when teenagers with ADHD (16-18) had their cars outfitted with on-board cameras facing the cabin and the roadway, there was no difference in rates of risky driving during the first and last weeks (Fabiano et al., 2016), and collaterals (parents) and teens illustrated coercive interactions strategies during these on-board assessments (Schatz, Fabiano et al., 2014). In addition, parenting and teen behaviors in the laboratory regarding a conflictual topic yielded sufficient behavioral variability across positive and negative parent/teen behaviors (Fabiano et al., 2016); it is expected that in-home, ecological, momentary assessment will be even more effective at generating information on social functioning. These results suggest that there will be acceptable rates of behavioral variability during the two-week assessment period and this is also an assessment period of reasonable length to prevent attrition.

ELIGIBILITY:
Inclusion Criteria:

All participants will have an estimated IQ greater than 70, a valid driving license/permit, and no evidence of psychosis or autism spectrum disorder at level 2 or 3. Individuals will be classified in the ADHD group if they meet DSM-5 criteria for ADHD based on the evaluation. Individuals who do not meet criteria for ADHD will be placed in the non-ADHD group.

Exclusion Criteria:

Medication use for ADHD will be an exclusion criteria, unless the participant works with the prescribing physician to take a 2-week holiday from medication for the duration of the study.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be between 16-30 years of age and have an identified collateral rater (e.g., parent, partner). Half of the participants will have ADHD and the other half will not meet diagnostic criteria for ADHD. To reduce variability between the ADHD and non-ADHD groups, we will match participants on age (+/- 2 years), sex, and whether they are employed or unemployed.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Social Impairment | 14 days
  Ecological, momentary assessment of social interaction impairment
ADHD symptoms | 14 days
  Ecological, momentary assessment of ADHD symptoms
Driving behavior | 14 days
  Sum of risky driving events (e.g., texting while driving; hard braking or acceleration
Percent of Behavioral Goals Met | 14 days
  Percent of daily schedule goals met on time

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Fabiano, Principal Investigator — Florida International University
Locations (1):
- Center for Children and Families, Amherst, New York, United States

IPD SHARING:
Plan to Share IPD: No